CLINICAL TRIAL: NCT07229937
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Dose-ranging Study to Evaluate the Efficacy and Safety of HRS-1301 in Participants With Dyslipidemia
Brief Title: A Phase II Study To Evaluate the Efficacy And Safety Of HRS-1301 In Participants With Dyslipidemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shandong Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS-1301-201
Record Dates: First submitted 2025-11-14; First posted 2025-11-17 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-09

CONDITIONS: Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- HRS-1301 Group A (Experimental)
  Interventions: Drug: HRS-1301
- HRS-1301 Group B (Experimental)
  Interventions: Drug: HRS-1301
- HRS-1301 Group C (Experimental)
  Interventions: Drug: HRS-1301
- HRS-1301 Group D (Experimental)
  Interventions: Drug: HRS-1301
- HRS-1301 Group E (Experimental)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HRS-1301 — HRS-1301 Dose 1，oral
  Arms: HRS-1301 Group A
Drug: HRS-1301 — HRS-1301 Dose 2，oral
  Arms: HRS-1301 Group B
Drug: HRS-1301 — HRS-1301 Dose 3，oral
  Arms: HRS-1301 Group C
Drug: HRS-1301 — HRS-1301 Dose 4，oral
  Arms: HRS-1301 Group D
Drug: Placebo — Placebo，oral
  Arms: HRS-1301 Group E

SUMMARY:
The purpose of the study is to explore the reasonable dosage of HRS-1301 in participants with dyslipidemia. The efficacy and safety of HRS-1301 will be evaluated after 12-weeks treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female ≥ 18 years old, who is able and willing to provide a written informed consent
2. BMI ≥ 18.0 kg/m2
3. Clinically diagnosed with ASCVD and LDL-C ≥ 1.8 mmol/L OR, if no history of ASCVD, has intermediate to high risk of developing ASCVD and LDL-C ≥ 2.6 mmol/L
4. Male and female subjects of childbearing potential and their partners must have no plans to donate sperm or become pregnant during the entire study period and for 2 weeks after the last dose, and agree to use contraceptive methods as specified in the protocol

Exclusion Criteria:

1. TG > 5.6 mmol/L
2. Diagnosed with homozygous familial hypercholesterolemia (HoFH)
3. Acute ischemic ASCVD events within 12 months before screening, or during the screening and run-in phase
4. Heart failure with New York Heart Association (NYHA) Class III-IV
5. Malignant tumors within 5 years
6. Received or is regularly receiving LDL or plasma apheresis within 12 months before screening
7. History or presence of severe gastrointestinal, hepatic, or renal diseases, or other known diseases that may interfere with drug absorption, distribution, metabolism, or excretion
8. Uncontrolled diabetes mellitus and/or hypertension
9. Has undergone transplantation of any vital organ, such as lung, liver, heart, bone marrow, or kidney

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Estimated)
Dates: Start 2025-11-25 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Percentage change in LDL-C relative to baseline | at 12 weeks of treatment

SECONDARY OUTCOMES:
Proportion of subjects achieving LDL-C goals | at 12 weeks of treatment
Percentage change in TC relative to baseline； | at 12 weeks of treatment
Percentage change in HDL-C relative to baseline； | at 12 weeks of treatment
Percentage change in TG relative to baseline； | at 12 weeks of treatment
Percentage change in non-HDL-C relative to baseline； | at 12 weeks of treatment
Percentage change in ApoB relative to baseline； | at 12 weeks of treatment
Percentage change in ApoA1 relative to baseline； | at 12 weeks of treatment；
Percentage change in Lp(a) relative to baseline； | at 12 weeks of treatment；
Percentage change in hsCRP relative to baseline； | at 12 weeks of treatment；
Number of participants with one or more adverse events | during the study period；Approximately half a year

CONTACTS AND LOCATIONS:
Locations (1):
- The 2nd Affiliated Hospital of Harbin, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: Undecided